CLINICAL TRIAL: NCT00414661
Title: A Prospective Observational Study To Evaluate Long-Term Safety And Functional Status Of Subjects With Rheumatoid Arthritis Previously Enrolled In Studies Of CP-690,550
Brief Title: Long-Term Safety Follow-Up Of Subjects Previously Enrolled In Rheumatoid Arthritis Studies Of CP-690,550
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921029
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Observational non-interventional long-term safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: All enrolled subjects
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Subjects had to have received CP-690,550 or other blinded study drug in index study. No intervention in this long-term follow-up trial.

SUMMARY:
The purpose of this study is to follow the health of subjects who have previously been enrolled in studies of CP-690,550 for treatment of their rheumatoid arthritis. Subjects are only eligible for this study after they have completed all participation in other studies of CP-690,550.

DETAILED DESCRIPTION:
At their last visit of a qualifying study, eligible subjects will be given the opportunity to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed all participation in any other Phase 2B or Phase 3 studies of CP-690,550 for rheumatoid arthritis.

Exclusion Criteria:

* Any subject who refuses consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received at least one dose of study drug and ceased participation in any Phase 2B or 3 randomized, controlled or open-label (qualifying) study of CP-690,550 for the treatment of RA, but are no longer receiving CP-690,550.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2007-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (18):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Tacoma, Washington
- Pfizer Investigational Site, Buenos Aires, Argentina
- Brazil (3):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Sofia, Bulgaria
- Pfizer Investigational Site, Victoria, British Columbia, Canada
- Chile (2):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 11 - Chodov
- Pfizer Investigational Site, Santo Domingo, Santo Domingo Province, Dominican Republic
- Pfizer Investigational Site, Hyvinkää, Finland
- Greece (2):
  - Pfizer Investigational Site, Athens, Goudi
  - Pfizer Investigational Site, Thessaloniki
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Szolnok
  - Pfizer Investigational Site, Veszprém
- India (3):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
- Italy (2):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Genova
- Japan (4):
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Higashihiroshima, Hiroshima
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo
- Mexico (2):
  - Pfizer Investigational Site, México, D.f.
  - Pfizer Investigational Site, Mexico City, Mexico City
- Poland (5):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, San Juan, Puerto Rico
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Žilina
- South Korea (4):
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
- Pfizer Investigational Site, Guadalajara, Guadalajara, Spain
- Pfizer Investigational Site, Vinnitsa, Ukraine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921029&StudyName=Long-Term%20Safety%20Follow-Up%20Of%20Subjects%20Previously%20Enrolled%20In%20Rheumatoid%20Arthritis%20Studies%20Of%20CP-690%2C550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received at least 1 dose of CP-690,550, placebo or adalimumab for the treatment of Rheumatoid Arthritis (RA) in previous studies and had ceased participation in other Phase 2B or 3 randomized, controlled or open-label study of CP-690,550 were eligible for this study.
Groups:
- CP-690,550 >=10 mg: Participants who had received 1 dose CP-690,550 greater than or equal to (>=) 10 milligram (mg) orally twice daily in any of the previous studies.
- CP-690,550 <10 mg: Participants who had received 1 dose CP-690,550 less than (<) 10 mg orally twice daily in any of the previous studies.
- Placebo: Participants who had received 1 dose of matching-placebo in any of the previous studies.
- Adalimumab: Participants who had received 1 dose of adalimumab in any of the previous studies.
Period: Overall Study
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Started | 48 | 89 | 22 | 3
Completed | 34 | 75 | 20 | 0
Not Completed | 14 | 14 | 2 | 3
Not completed — Death | 2 | 5 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 2 | 2
Not completed — Other | 6 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab | Total
Number analyzed (Participants) | 48 | 89 | 22 | 3 | 162
Age Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.8) | 54.7 (11.6) | 51.8 (13.5) | 52.3 (16.0) | 55.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 72 | 17 | 3 | 132
  Male | 8 | 17 | 5 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Lymphoproliferative Disorders (LPD)
Description: Incidence rate was calculated separately for active treatment period and follow-up period in previous studies as number of participants with LPD by number of days while on active treatment or during follow-up period per 100 person-years. Standardization of incidence rates was based upon the age and sex distribution of the entire study population.
Time Frame: Up to Month 24
Population: Safety analysis set included all participants who were previously enrolled in either randomized, controlled or open-label studies of CP-690,550 and had signed the informed consent form for this study.
Measure: Number (95% Confidence Interval); unit: LPD per 100 person-years
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 48 | 89 | 22 | 3
LPD per 100 person-years | NA [NA to NA] — Data was not analyzed as no LPD occurred. | NA [NA to NA] — Data was not analyzed as no LPD occurred. | NA [NA to NA] — Data was not analyzed as no LPD occurred. | NA [NA to NA] — Data was not analyzed as no LPD occurred.

2. Primary Outcome: Incidence of Lymphoma
Description: Incidence rate was calculated separately for active treatment period and follow-up period in previous studies as number of participants with lymphoma by number of days while on active treatment or during follow-up period per 100 person-years. Standardization of incidence rates was based upon the age and sex distribution of the entire study population.
Time Frame: Up to Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Lymphoma per 100 person-years
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 48 | 89 | 22 | 3
Lymphoma per 100 person-years | NA [NA to NA] — Data was not analyzed as no lymphoma occurred. | NA [NA to NA] — Data was not analyzed as no lymphoma occurred. | NA [NA to NA] — Data was not analyzed as no lymphoma occurred. | NA [NA to NA] — Data was not analyzed as no lymphoma occurred.

3. Primary Outcome: Incidence of Important Infections
Description: Incidence rate was calculated separately for active treatment period and follow-up period in previous studies as number of participants with important infections by number of days while on active treatment or during follow-up period per 100 person-years. Standardization of incidence rates was based upon the age and sex distribution of the entire study population.
Time Frame: Up to Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Infections per 100 person-years
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 48 | 89 | 22 | 3
Infections per 100 person-years | 0.000 [0.000 to NA] — Upper limit of 95 percent (%) confidence interval (CI) was not estimable as no event occurred in this arm group. | 0.607 [0.086 to 4.312] | 0.000 [0.000 to NA] — Upper limit of 95 percent (%) confidence interval (CI) was not estimable as no event occurred in this arm group. | 0.000 [0.000 to NA] — Upper limit of 95 percent (%) confidence interval (CI) was not estimable as no event occurred in this arm group.

4. Other Pre Specified Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: Safety analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for the measure and 'n' signifies participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 48 | 88 | 22 | 3
units on a scale
  Baseline (n= 48, 88, 22, 3) | 1.32 (0.67) | 1.42 (0.67) | 1.63 (0.76) | 1.13 (0.13)
  Month 6 (n= 37, 81, 21, 2) | 1.08 (0.61) | 1.23 (0.69) | 1.21 (0.82) | 0.19 (0.27)
  Month 12 (n= 39, 79, 21, 1) | 1.16 (0.63) | 1.12 (0.76) | 1.15 (0.81) | 0.88 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Month 18 (n= 35, 76, 20, 0) | 1.15 (0.59) | 1.07 (0.77) | 1.12 (0.86) | NA (NA) — Data was not analyzed as no participants were evaluable in this arm group.
  Month 24 (n= 31, 68, 20, 0) | 1.15 (0.69) | 1.14 (0.78) | 1.07 (0.87) | NA (NA) — Data was not analyzed as no participants were evaluable in this arm group.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 >=10 mg | CP-690,550 <10 mg | Placebo | Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/89 | 0/22 | 0/3
Other Adverse Events (participants affected / at risk) | 3/48 | 2/89 | 1/22 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 >=10 mg (N=48) | CP-690,550 <10 mg (N=89) | Placebo (N=22) | Adalimumab (N=3)
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 >=10 mg (N=48) | CP-690,550 <10 mg (N=89) | Placebo (N=22) | Adalimumab (N=3)
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.